CLINICAL TRIAL: NCT06533059
Title: AKTive-001: A Phase 1/1b Multiple Cohort Trial of ALTA2618 in Patients With Advanced Solid Tumors With AKT1 E17K Mutation
Brief Title: A Study to Learn About Study Medicine ALTA2618 in Adults With AKT1 E17K-Mutant Solid Tumors
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Alterome Therapeutics, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2618-001
Record Dates: First submitted 2024-07-25; First posted 2024-08-01 (Actual); Last update posted 2025-11-26 (Actual); Status verified 2025-02

CONDITIONS: Cancer; Breast Cancer; Endometrial Cancer; Metastatic Cancer; Advanced Solid Tumor
Keywords: AKT1 E17K; Breast cancer; Breast carcinoma; Breast neoplasm; ER positive breast; HR positive breast; Triple negative breast cancer; Gynecologic cancer; Gynecologic neoplasm; Gynecologic carcinoma; Endometrial cancer; Endometrial neoplasm; Endometrial carcinoma; Cervical cancer; Cervical neoplasm; Cervical carcinoma; Ovarian cancer; Ovarian carcinoma; Ovarian neoplasm; Fallopian cancer; Fallopian carcinoma; Fallopian neoplasm; Prostate cancer; Prostate carcinoma; Prostate neoplasm; Solid tumors; AKT mutation; Mutant AKT; AKT1 mutation; AKT mutant; AKT1E17K
MeSH Terms: conditions — Neoplasms; Breast Neoplasms; Endometrial Neoplasms; Neoplasm Metastasis; Triple Negative Breast Neoplasms; Genital Neoplasms, Female; Uterine Cervical Neoplasms; Ovarian Neoplasms; Prostatic Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- ALTA2618 (Experimental): ALTA2618 will be administered continuously at a protocol-defined dose based on cohort assignment
  Interventions: Drug: ALTA2618

INTERVENTIONS:
Drug: ALTA2618 — Oral ALTA2618 tablets will be administered at protocol-defined dose

SUMMARY:
The purpose of this study is to characterize the safety and tolerability of ALTA2618 in adults with AKT1 E17K-mutant advanced solid tumors.

DETAILED DESCRIPTION:
This is an open-label, multicenter, Phase 1/1b study of ALTA2618, a mutant-selective and orally bioavailable AKT1 E17K inhibitor, in adults with AKT1 E17K-mutant solid tumors. This study will evaluate the safety, tolerability, pharmacokinetics (PK), and preliminary clinical activity of ALTA2618, and aims to find the best dose. The study consists of two parts: Part 1 - Dose Escalation and Part 1b - Dose Expansion.

ELIGIBILITY:
Inclusion Criteria:

* Histologically confirmed diagnosis of a solid tumor malignancy harboring AKT1 E17K mutation identified through molecular testing (NGS- or PCR-based) with a Clinical Laboratory Improvement Amendments-certified (or equivalent) diagnostic test.
* Unresectable or metastatic disease
* Progressed on, intolerant to, or declined prior standard-of-care therapy (including targeted therapy, if applicable) appropriate to tumor type and stage
* Evaluable or measurable disease per RECIST v1.1
* Eastern Cooperative Oncology Group (ECOG) performance status of 0 or 1.
* Adequate organ function.

Exclusion Criteria:

* Prior treatment with PI3K and/or mTOR inhibitors
* Patients known to have KRAS, NRAS, HRAS, or BRAF genomic alterations in their tumor
* Known condition that prohibits ability to swallow or absorb an oral medication

Other inclusion/exclusion criteria may apply.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 110 (Estimated)
Dates: Start 2024-08-22 (Actual); Primary Completion 2026-12-29 (Estimated); Study Completion 2027-12-29 (Estimated)

PRIMARY OUTCOMES:
Adverse Events | Up to 39 months
  Number of participants that experience treatment-emergent adverse events (TEAEs).
Dose Limiting Toxicities | 21 days
  Number of participants with Dose Limiting Toxicities (DLTs).

SECONDARY OUTCOMES:
Maximum Observed Plasma Concentration (Cmax) | Cycle 1 (each cycle is 21 days) Day 1 (or Lead-in) and Day 8: Predose and up to 24 hours postdose
  Cmax
Time to Reach Maximum Observed Plasma Concentration (Tmax) | Cycle 1 (each cycle is 21 days) Day 1 (or Lead-in) and Day 8: Predose and up to 24 hours postdose
  Tmax
Area Under Plasma Concentration Time Curve During the Dosing Interval (AUCt) | Cycle 1 (each cycle is 21 days) Day 1 (or Lead-in) and Day 8: Predose and up to 24 hours postdose
  AUCt
Terminal Half-Life (t1/2) | Cycle 1 (each cycle is 21 days) Lead-in phase: Predose and up to 72 hours postdose
  t1/2
Overall Response Rate (ORR) | Up to 39 months
  Assess per RECIST 1.1
Duration of Response (DOR) | Up to 39 months
  Assess per RECIST 1.1
Progression-Free Survival (PFS) | Up to 39 months
  Assess per RECIST 1.1
Overall Survival (OS) | Up to 39 months
  Assess per RECIST 1.1

CONTACTS AND LOCATIONS:
Overall Officials: Study Medical Director, Study Director — Alterome Therapeutics
Locations (40):
- United States (17):
  - Research Site, La Jolla, California
  - Research Site, Los Angeles, California
  - Research Site, Denver, Colorado
  - Research Site, Sarasota, Florida
  - Research Site, Atlanta, Georgia
  - Research Site, Boston, Massachusetts
  - Research Site, St Louis, Missouri
  - Research Site, Mineola, New York
  - Research Site, New York, New York
  - Research Site, Maumee, Ohio
  - Research Site, Nashville, Tennessee
  - Research Site, Dallas, Texas
  - Research Site, Houston, Texas
  - Research Site #2, San Antonio, Texas
  - Research Site, San Antonio, Texas
  - Research Site, Fairfax, Virginia
  - Research Site, Madison, Wisconsin
- Australia (5):
  - Research Site, Blacktown, New South Wales
  - Research Site, Randwick, New South Wales
  - Research Site, South Brisbane, Queensland
  - Research Site, Malvern, Victoria
  - Research Site, Nedlands, Western Australia
- France (4):
  - Research Site, Caen
  - Research Site, Dijon
  - Research Site, Saint-Herblain
  - Research Site, Villejuif
- Japan (4):
  - Research Site, Kyoto
  - Research Site, Matsuyama
  - Research Site, Shizuoka
  - Research Site, Tokyo
- Research Site, Seoul, South Korea
- Spain (3):
  - Research Site, Barcelona
  - Research Site, Madrid
  - Research Site, Valencia
- Taiwan (2):
  - Research Site, Changhua
  - Research Site, Taipei
- United Kingdom (4):
  - Research Site, London
  - Research Site, Manchester
  - Research Site, Newcastle upon Tyne
  - Research Site, Sutton